CLINICAL TRIAL: NCT03765658
Title: An Ascending Single-Dose Safety, Tolerability and Exposure Study to Explore the Maximum Tolerated Dose of GRT0151Y in Healthy Adult Non-dependent Recreational Opiate Users
Brief Title: A Clinical Study in Healthy Adults Who Sometimes Take Drugs for Pleasure to Investigate the Safety and Tolerability of GRT0151Y and to Find Out Which Single Dose of the Compound is Maximally Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HP0151Y/10; PK872A (Other: Sponsor)
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Pain; Acute Pain; Chronic Pain
MeSH Terms: conditions — Pain; Acute Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: During each treatment period, participants randomly received either GRT0151Y or matching placebo, in a manner that no participant received placebo in two consecutive periods.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GRT0151Y dose escalation (Experimental): GRT0151Y will be administered to participants as 50 mg capsules in a dose escalation range of 150, 200, 250, 300, 350 and 400 mg. Dose levels were increased by increments of 50 mg to a maximum of 400 mg, only after the previous dose level was found to be well-tolerated. During each treatment period, participants randomly received either GRT0151Y or matching placebo, in a manner that no participant received placebo in two consecutive periods.
  Interventions: Drug: GRT0151Y dose escalation; Drug: Matching placebo

INTERVENTIONS:
Drug: GRT0151Y dose escalation — Single doses of 150, 200, 250, 300, 350 and 400 mg (3, 4, 5, 6, 7 or 8 capsules of 50 mg)
Drug: Matching placebo — Matching placebo capsules (3, 4, 5, 6, 7 or 8 capsules)

SUMMARY:
The purpose of this study is to determine the maximum dose of GRT0151Y that is tolerable and to explore the safety profile of the drug.

For each Treatment Period (Visits 2-5), dosing will be separated by at least one week. Participants in this study will receive up to four doses of the study drug and up to two placebo (an inactive substance) preparations, one at a time on each of up to six visits. Participants will receive a single dose of either GRT0151Y or placebo beginning with the lowest dose of study drug 150 milligrams (mg), followed by 200 mg, 250 mg, 300 mg, 350 mg and 400 mg doses of the study drug. Participants will only be allowed to proceed to the next higher dose of GRT0151Y (or placebo) if the previous dose was well tolerated. Neither the participant nor the study staff will know whether participants are receiving GRT0151Y or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 55 years of age, inclusive.
* Acceptable body mass index (BMI) (weight [kilograms]/height (square meter) range of 19 to 30 kilograms per square meter, inclusive).
* Signed an informed consent document indicating that they understand the purpose of and procedures required for the study, and are willing to participate in the study.
* Participants with a history of recreational opiate use (defined as nontherapeutic use at least 10 times in the past year and at least once in the last 12 weeks prior to screening) but not dependent on opiates Diagnostic and Statistical Manual of Mental Disorders-4th edition (DSM-IV criteria).
* Participants must consent to use a medically acceptable method of contraception throughout the entire study period, including washout periods. For all females of childbearing potential only: adequate contraception is defined as any form of hormonal contraception or intra-uterine device that needs to be in place for a period of at least two months prior to screening. Additional barrier contraception must be used for the duration of the study, defined as from the time of the enrolment visit to the final examination, and for at least one full month thereafter. A single barrier method alone or abstinence alone is not acceptable. Women of non-childbearing potential may be included if surgically sterile or post-menopausal for at least two years.
* Female participants of childbearing potential must have a negative pregnancy test (beta- Human chorionic gonadotropin) at the enrolment visit. For females of childbearing potential, the time between the enrolment visit and first receipt of drug will be separated by a minimum of 10 days to ensure accuracy of the pregnancy test.
* Participants with a positive urine drug screen (for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, phencyclidine and opiates) upon presentation at enrolment will be allowed to continue only if the investigator or designee considers that the presence of the drug will not introduce additional risk factors for the study participant, or interfere with study procedures or data integrity. Positive drug screens for select drugs are to be confirmed using quantitative methods such as GC/MS or equivalent, and the investigator or designee's decision to allow participants to continue will take into account the quantitative levels of drug in the subjects' urine. Participants may be rescheduled for another treatment period at the investigator's discretion.
* Deemed healthy on the basis of enrolment visit physical examination, medical history, vital signs, and clinical laboratory parameters (serum/urine biochemistry, urinalysis, clotting, blood sedimentation rate (BSR), haematology and hepatitis and human immunodeficiency virus (HIV) virus serology). If the results of the laboratory tests or the urinalysis testing are not within the laboratory's reference ranges, the participant can be included only on condition that the investigator or designee judges that the deviations are not clinically relevant and do not interfere with the study objectives.
* Must have a negative breath alcohol analysis at enrolment. A positive alcohol reading is one that is above the error measurement associated with the breathalyzer. Participants presenting a positive alcohol breath test may be allowed to continue in the study only if the investigator (or designee) considers that the presence of breath alcohol does not suggest problematic alcohol consumption, and will not introduce additional risk factors for the study participant, or interfere with study procedures or data integrity.
* Ability to speak, read and understand English sufficiently to understand the nature of the study, to provide written informed consent and to allow completion of all study assessments.

Exclusion Criteria:

* History of or current substance dependence (except nicotine and caffeine dependence), as defined by the DSM-IV.
* Participants attempting to discontinue their recreational drug use, or who have been in a drug rehabilitation program in the 12 months prior to enrolment.
* History or risk of seizures (i.e. head trauma, epilepsy in family, anamnesis, unclear loss of consciousness).
* Positive HIV type 1/2 antibodies, hepatitis B surface (HBs) antigen, hepatitis B core (HBc) antibodies (Immunoglobulin and Immunoglobulin M), hepatitis C virus (HCV) antibodies.
* Participants with gastrointestinal disease (e.g., paralytic ileus) or constipation or who have clinically significant gastrointestinal problems, including narrowing (pathologic or iatrogenic) of the gastrointestinal tract, or other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Participants with a history of or current Chronic Obstructive Pulmonary Disease, or any other lung disease, (e.g., asthma, sleep apnea) that would cause carbon dioxide (CO2) retention.
* Participants with a history of or current cardiovascular dysfunction including marked repolarization abnormality (e.g., suspicious or definite congenital long QT syndrome, resting pulse rate between 45 or 95 beats per minute, and orthostatic or uncontrolled hypotension or hypertension (systolic blood pressure less than or equal to 100 and greater than or equal to 140 Millimeter mercury (mmHg), diastolic blood pressure less than or equal to 50 and greater than or equal to 95 mmHg), or use of co-medication that is known to influence cardiac repolarization substantially, evaluated at enrolment.
* QT/QTc values greater than 500 milliseconds at enrolment and/ or randomization.
* Male participants with hemoglobin less than 125 grams per Liter and female participants with hemoglobin less than 115 grams per Liter.
* Blood donation (more than 100 milliliter) or comparable blood losses within 30 days prior to the start of the study.
* Known contraindications/hypersensitivity to other opioids, naloxone, benzodiazepines, hydromorphone or definite or suspected allergy or hypersensitivity to drugs having a similar mechanism of action as the study drug.
* Pregnant or lactating.
* Participants who have used any prescription medication (except for sex-hormone replacement or birth control medications) including known CYP2D6 inhibitors and substrates which lower the seizure threshold within 14 days prior to the first study drug administration or monoamine-oxidase inhibitors (MAOIs) within 21 days prior to the first study drug administration.
* Participants who have used tricyclic antidepressants (TCA), selective serotonin re-uptake inhibitors (SSRI), selective norepinephrine reuptake inhibitors (SNRI), and antiparkinsonian drugs within 30 days prior to the first study drug administration.
* Participants who plan to take prescription medication, over-the-counter, or herbal medications while in the study, with the exception of birth control medications, sex-hormone replacement, vitamins/minerals and acetaminophen (up to 2 gram per day).
* Participants who have taken a new chemical entity under development within the last 30 days prior to receiving the first dose of IMP or longer, if on the basis of pharmacokinetic/pharmacodynamic characteristics, a possible interaction with study objective cannot be reasonably excluded.
* Not able to abstain from consuming caffeine containing beverages or foods (tea, coffee, chocolate or cola). Participants not able to refrain from smoking more than 20 cigarettes per day.
* Serum creatinine higher than 1.5 times the upper limit of normal range at enrolment.
* Any documented or suspected DSM-IV psychiatric disorder currently or within the past year, or any prior psychiatric condition that might compromise subject safety by increasing the risk of an untoward effect from the study drugs administered in this study as determined by the investigator's or designee's assessment of the Symptom Checklist 90-R (SCL-90-R) results.
* Participants who, in the investigator's opinion, may not be capable of following the study schedule for any reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2006-01-20 (Actual); Primary Completion 2006-03-02 (Actual); Study Completion 2006-03-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of GRT0151Y | First dose to Last dose assessed to be well tolerated. From Day 1 to Day 3 (for up to 6 periods)
  The progression to the next higher dose group occurred only after a thorough risk-benefit assessment, based upon the safety and tolerability data of the participants from the completed trial group (interim safety report [ISR]). The ISRs were prepared by the investigator and were submitted to the sponsor for benefit-risk assessment. The MTD would have been reached if the benefit-risk assessment had been unfavorable to progress to the next higher dose group.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GRT0151Y | pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 32 and 48 hours post dose
  Blood samples were obtained and plasma concentrations were determined using a validated stereoselective liquid chromatography-tandem mass spectrometry (LC-MS/MS).
Time to reach maximum plasma concentration (tmax) of GRT0151Y | pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 32 and 48 hours post dose
  Blood samples were obtained and plasma concentrations were determined using a validated stereoselective LC-MS/MS.
Area under the plasma concentration-time curve (AUC0-t) | pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 32 and 48 hours post dose
  Blood samples were obtained and plasma concentrations were determined using a validated stereoselective LC-MS/MS.
Divided Attention Test (DAT) | pre-dose, and 1, 2, 4, 6, 8, 12, 24, 32 and 48 hours post-dose
  Manual-tracking test with a simultaneous visual target detection component. Participant is provided with joystick and presented with the image of an airplane and a randomly curving road; participant has to position the airplane over the center of the road while being distracted repeatedly by visual targets they have to respond to. Percentage of time over the road (milliseconds), response latency of correct responses and percentage of target hits are recorded.
Choice Reaction Time (CRT) | pre-dose, and 1, 2, 4, 6, 8, 12, 24, 32 and 48 hours post-dose
  Choice reaction time (CRT) is a computerized assessment that trains the participant to respond to stimuli presented on the screen. The task requires the participant to react as soon as a colored key appears in one of up to eight locations. The participant must respond by lifting their finger from the central start button and depressing the corresponding response key as quickly as possible. This is the reaction time (RT). Lower scores indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Ventana Clinical Research Corporation, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No